CLINICAL TRIAL: NCT01961804
Title: Phase 3 Study Comparing Preventive Reversal of Vitamine K Antagonist Versus Reversion Only in Case of Intracranial Bleeding in Patients Receiving Vitamine K Antagonist Treatment
Brief Title: PREVACT : Preventive REversal of Vitamine K Antagonist in Minor Craniocerebral Trauma
Acronym: PREVACT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRC 2012-02
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Last update posted 2021-04-27 (Actual); Status verified 2020-08

CONDITIONS: Coagulation; Intravascular; Craniocerebral Trauma; Haemorrhage
MeSH Terms: conditions — Thrombosis; Craniocerebral Trauma; Hemorrhage

ARMS (2):
- Actual recommendations (Other): Current guidelines recommend to perform a CT scan and realise the anticoagulation reversion only in case of intracranial bleeding diagnosed.
  Interventions: Drug: Reversion
- Preventive reversion (Experimental): Realise a preventive reversion before performing any CT scan.
  Interventions: Drug: Reversion

INTERVENTIONS:
Drug: Reversion — Administration of prothrombin complex concentrates: KANOKAD before CT Scan
  Other Names: KANOKAD

SUMMARY:
The occurence of a minor craniocerebral trauma in patients receiving vitamine K antagonist treatment leads to a high risk of bleeding.

Current guidelines recommend to perform a CT scan, and, in case of intracranial bleeding, to reverse anticoagulation with concomitant administration of prothrombin complex concentrates (PCCs) and vitamin K.

However, even if a reversion is performed, the prognostic of post-traumatic intracranial bleeding remain bad.

The investigators hypothesize that, for patients admitted in an emergency department after a minor head trauma and receiving anticoagulant treatment, a systematic preventive reversion with PCCs can lead to a significant reduction of intracranial haemorrhage and can also improve the neurological prognostic of patients versus the current strategy.

PREVACT will test this hypothesis, in an open label, randomized, multicentre, clinical trial involving 400 patients.

ELIGIBILITY:
Inclusion Criteria:

* Admission in an emergency departement for a recent and isolated minor head trauma with at least one of the following characteristic : a period of alteration in the level of consciousness, a period of loss of consciousness (< 30 min), a posttraumatic amnesia, persistant posttraumatic headache, repeated vomitting (at least 2 episodes) or any other neurological sign such a convulsion or a localised neurological sign, wound of the scalp or the face testifying of the importance of the cranial trauma...
* Subject receiving anticoagulant treatment with anti-vitamin K for the treatment of atrial fibrillation (AF)
* Initial ED Glasgow Coma Scale (GCS) score of ≥13
* Achievable follow up
* Informed consent form signed by the patient or if he/she isn't able an emergency inclusion can be realised.

Exclusion Criteria:

* Delay between the minor head trauma and the possible preventive PCC's administration > 6h
* Subject receiving anticoagulant treatment other than anti vitamin K (heparin, fondaparinux, dabigatran, rivaroxaban, apixaban...)
* Subject receiving anticoagulant treatment for other reason than a AF
* Subject on antiplatelet treatment (except the use of low dose of aspirin (≤ 100 mg/day)
* Delocalised biology INR in capillary blood < 1.5 if it's available (only in departement where this analyse is a usual practice)
* Haemorrhage or suspected haemorrhage other than intracranial which could led to a reversion of the anticoagulation
* Head trauma associated with one or further potential haemorrhagic traumatic lesions
* Subject who reject the use of products derived from human blood
* Women who are pregnant
* Subject with any condition that, as judged by the investigator, would place the subject at increased risk of harm if he/she participated in the study
* Subject without social security registered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-09-03 (Actual)

PRIMARY OUTCOMES:
Percentage of intracranial bleeding diagnosed in CT scan | 24 hours +/- 4 hours
  This primary outcome measure will be analyse in a centralised place by two neuro-radiologist in blind of the randomised group.

SECONDARY OUTCOMES:
Volumetric measure of intracranial haemorrhage | CT scan performed 24 hours +/-4 after inclusion
  This secondary outcome measure will be analyse in a centralised place by two neuro-radiologist in blind of the randomised group.
Percentage of patient having a decrease in their autonomy | 3 months
  A loss of at least one point in the Glasgow Outcome Score Extended
Percentage of patient having a systemic or neurologic ischemic attacks | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: ROY Pierre-Marie, Professor, Principal Investigator — UH Angers; TAZAROURTE Karim, Pr, Study Chair — UH Lyon
Locations (21):
- France (21):
  - CH Agen, Agen
  - CHU Angers, Angers
  - Ch Annecy, Annecy
  - CHU Chateauroux, Châteauroux
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CHG du Mans, Le Mans
  - Ch Les Sables D'Olonne, Les Sables-d'Olonne
  - Ch Longjumeau, Longjumeau
  - HCL Edouard Herriot, Lyon
  - CHU METZ, Metz
  - Chg Montauban, Montauban
  - Chu Nantes, Nantes
  - CHU Nice, Nice
  - CHU Pitié Salpétrière, Paris
  - Chu Tenon, Paris
  - Chu Poitiers, Poitiers
  - Chu Saint Brieuc, Saint-Brieuc
  - Ch Saint Malo, St-Malo
  - Chu Toulouse, Toulouse
  - Chu Tours, Tours
  - Ch Versailles, Versailles

REFERENCES:
- [Derived] Douillet D, Tazarourte K, Dehours E, Brice C, Andrianjafy H, Trinh-Duc A, Lasocki S, Labriffe M, Riou J, Roy PM. Systematic vitamin K antagonist reversal with prothrombin complex concentrate in patients with mild traumatic brain injury: randomized controlled trial. Eur J Emerg Med. 2025 Jun 1;32(3):180-187. doi: 10.1097/MEJ.0000000000001199. Epub 2024 Nov 6. PMID 40315031